CLINICAL TRIAL: NCT01765530
Title: Endotracheal Tubes Cleaned With a Novel Mechanism for Secretions Removal
Brief Title: Efficacy Study of a Novel Device to Clean the Endotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: West Virginia University (Other); endOclear, LLC. (Unknown)
Responsible Party: Principal Investigator, Robert M. Kacmarek, Director, Respiratory Care Services; Professor of Anesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MGH-ETT cleaning
Record Dates: First submitted 2012-12-28; First posted 2013-01-10 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-04

CONDITIONS: Endotracheal Extubation; Airway Obstruction; Airway Control; Pneumonia, Ventilator-Associated; Breathing Mechanics
Keywords: Medical Devices; Ventilator-Associated Pneumonia (VAP); Ventilator-Associated Events (VAE); Endotracheal Tube; Microbial Diversity; Anti-Resistance; Computed Tomography (CT)
MeSH Terms: conditions — Airway Obstruction; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETT cleaning manuver (Experimental): Patients randomized to the treatment group will undergo an ETT cleaning maneuver with endOclear three times a day (every 8 hours) for the whole intubation period in addition to the standard of care.
  Interventions: Device: ETT cleaning maneuver
- Standard of care (No Intervention): In the protocol no intervention is planned for the control group, which will therefore be treated with blind suctioning as per caregiver clinical decision.

INTERVENTIONS:
Device: ETT cleaning maneuver — EndOclear device will be used for ETT cleaning maneuver. This is a commercially available device. It consists of an ETT cleaning apparatus with a flexible central tube and a cleaning device at its distal end. The cleaning device has a mechanically expandable mesh structure which can be adapted to selectively move between a radially-collapsed position and a radially-expanded one. In operation, the collapsed cleaning apparatus is inserted into the ETT through a Y-shaped connector. The device is then expanded by a safety toggle protected trigger mechanism that, when fired, presses the device's smooth silicone disc against the inside surface of the ETT. The cleaning apparatus is then pulled out of the ETT removing mucus deposits and secretions.
  We will add endOclear to the standard ICU practice, scheduling the systematic use of the device every 8 hours for the whole intubation period.
  Arms: ETT cleaning manuver

SUMMARY:
The purpose of this study is to evaluate the in-vivo efficacy of a novel device (endOclear) for cleaning the endotracheal tube (ETT) lumen from secretions. The investigators hypothesize that a protocol of routine ETT cleaning with endOclear may increase the ETT luminal volume measured at extubation compared to the current standard of care. The device may therefore be clinically useful by better maintaining the ETT original function.

DETAILED DESCRIPTION:
After a few days of mechanical ventilation (MV), the lumen of the endotracheal tube (ETT) is coated with a thick bacterial biofilm, which is a potential source for bacterial colonization of the lower respiratory tract and ventilator-associated pneumonia (VAP). Accumulation of mucus/secretions on the interior of the ETT also effectively lowers the cross section of the ETT and increases significantly the work of breathing in intubated patients, who then require increased MV support, with prolonged intubation and ICU stay.

A primary goal for all ICUs is to shorten the time of MV, to decrease the incidence of ETT microbial colonization and ultimately VAP incidence. To meet this goal several airways technologies to maintain the ETT free from debris/bacteria have been developed in order to improve the current ventilator-liberation standards in intubated critically ill patients.

Based on preliminary laboratory, animal and clinical data, The investigators now wish to test the hypothesis that a novel commercially available ETT cleaning device can be effective in targeting two specific issues:

* Specific aim 1: To evaluate the mean difference in ETT luminal volume of ETTs cleaned with the novel cleaning device (EndOclear) vs. ETT cleaned in the standard manner.
* Specific aim 2: To determine whether ETTs cleaned with the novel device show a lower degree of microbial colonization for the entire period of mechanical ventilation.

Data about in-vivo respiratory mechanics measurements, microbial diversity and antibiotic resistance analysis, users' feedbacks and safety of the device will also be collected.

The investigators will conduct a clinical trial on 74 intubated patients randomized to receive standard ETT cleaning or cleaning with the EndOclear.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients expected to be intubated for at least 48 hours or longer
* Enrollment within 24 hours from intubation time

Exclusion Criteria:

* Current and past participation in another intervention trial conflicting with the present study
* Pregnant women and prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kacmarek, PhD, RRT, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Adair CG, Gorman SP, Feron BM, Byers LM, Jones DS, Goldsmith CE, Moore JE, Kerr JR, Curran MD, Hogg G, Webb CH, McCarthy GJ, Milligan KR. Implications of endotracheal tube biofilm for ventilator-associated pneumonia. Intensive Care Med. 1999 Oct;25(10):1072-6. doi: 10.1007/s001340051014. PMID 10551961
- [Background] Shapiro M, Wilson RK, Casar G, Bloom K, Teague RB. Work of breathing through different sized endotracheal tubes. Crit Care Med. 1986 Dec;14(12):1028-31. doi: 10.1097/00003246-198612000-00007. PMID 3780244
- [Background] Heyer L, Louis B, Isabey D, Lofaso F, Brochard L, Fredberg JJ, Harf A. Noninvasive estimate of work of breathing due to the endotracheal tube. Anesthesiology. 1996 Dec;85(6):1324-33. doi: 10.1097/00000542-199612000-00013. PMID 8968179
- [Background] Glass C, Grap MJ, Sessler CN. Endotracheal tube narrowing after closed-system suctioning: prevalence and risk factors. Am J Crit Care. 1999 Mar;8(2):93-100. PMID 10071699
- [Background] Shah C, Kollef MH. Endotracheal tube intraluminal volume loss among mechanically ventilated patients. Crit Care Med. 2004 Jan;32(1):120-5. doi: 10.1097/01.CCM.0000104205.96219.D6. PMID 14707569
- [Background] Boque MC, Gualis B, Sandiumenge A, Rello J. Endotracheal tube intraluminal diameter narrowing after mechanical ventilation: use of acoustic reflectometry. Intensive Care Med. 2004 Dec;30(12):2204-9. doi: 10.1007/s00134-004-2465-4. Epub 2004 Oct 2. PMID 15580475
- [Background] Villafane MC, Cinnella G, Lofaso F, Isabey D, Harf A, Lemaire F, Brochard L. Gradual reduction of endotracheal tube diameter during mechanical ventilation via different humidification devices. Anesthesiology. 1996 Dec;85(6):1341-9. doi: 10.1097/00000542-199612000-00015. PMID 8968181
- [Background] Berra L, Coppadoro A, Bittner EA, Kolobow T, Laquerriere P, Pohlmann JR, Bramati S, Moss J, Pesenti A. A clinical assessment of the Mucus Shaver: a device to keep the endotracheal tube free from secretions. Crit Care Med. 2012 Jan;40(1):119-24. doi: 10.1097/CCM.0b013e31822e9fe3. PMID 21926595
- [Background] Stone RH, Bricknell SS. Experience with a new device for clearing mucus from the endotracheal tube. Respir Care. 2011 Apr;56(4):520-2. doi: 10.4187/respcare.00642. Epub 2011 Jan 21. PMID 21255488
- [Background] Inglis TJ, Millar MR, Jones JG, Robinson DA. Tracheal tube biofilm as a source of bacterial colonization of the lung. J Clin Microbiol. 1989 Sep;27(9):2014-8. doi: 10.1128/jcm.27.9.2014-2018.1989. PMID 2778064
- [Background] Wilson AM, Gray DM, Thomas JG. Increases in endotracheal tube resistance are unpredictable relative to duration of intubation. Chest. 2009 Oct;136(4):1006-1013. doi: 10.1378/chest.08-1938. Epub 2009 May 1. PMID 19411293
- [Background] Berra L, Curto F, Li Bassi G, Laquerriere P, Baccarelli A, Kolobow T. Antibacterial-coated tracheal tubes cleaned with the Mucus Shaver : a novel method to retain long-term bactericidal activity of coated tracheal tubes. Intensive Care Med. 2006 Jun;32(6):888-93. doi: 10.1007/s00134-006-0125-6. Epub 2006 Apr 19. PMID 16601964
- [Background] Kolobow T, Berra L, Li Bassi G, Curto F. Novel system for complete removal of secretions within the endotracheal tube: the Mucus Shaver. Anesthesiology. 2005 May;102(5):1063-5. doi: 10.1097/00000542-200505000-00028. No abstract available. PMID 15851896

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ETT Cleaning Manuver | Standard of Care
Started | 37 | 37
Completed | 36 | 36
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETT Cleaning Manuver | Standard of Care | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (19) | 64 (17) | 62 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Occlusion Assessed Using a High Definition Computed Tomography Imaging of the Extubated ETTs
Description: The investigators will measure percentage of occlusion determined by the accumulation of secretion within the lumen of each ETT using a high definition Computed Tomography (CT) imaging of the extubated ETTs. The whole ETT will be analyzed through high-definition CT slices. 100% of occlusion means total occlusion of the lumen of the ETT and 0% means absence of any occlusion.
Time Frame: At extubation (An expected average of 5 days)
Measure: Mean (Standard Deviation); unit: percentage of occlusion
Arm/Group | ETT Cleaning Manuver | Standard of Care
Number analyzed (Participants) | 36 | 36
percentage of occlusion | 10.6 (8.0) | 17.7 (13.4)

2. Secondary Outcome: ETT Microbiology
Description: For each patient a quantitative culture will be obtained from the ETT after extubation. Secretions will be retrieved from the ETT after CT scan and quantitative standard cultures will be performed. Microbial molecular diversity analysis and antibacterial resistance patterns will also be studied.
Time Frame: At extubation (An expected average of 5 days)
Measure: Mean (Standard Error); unit: Log colony form unit (CFU)/ mL
Arm/Group | ETT Cleaning Manuver | Standard of Care
Number analyzed (Participants) | 36 | 36
Log colony form unit (CFU)/ mL | 2.89 (0.49) | 3.35 (0.48)

ADVERSE EVENTS:
Time Frame: Entire study 6 months
Arm/Group | ETT Cleaning Manuver | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes